CLINICAL TRIAL: NCT02183376
Title: Pharmacokinetics and Pharmacodynamics of BI 1356 5 mg Once Daily in Male and Female Subjects With Different Degrees of Liver Impairment (Child Pugh Classification A-C) as Compared to Male and Female Healthy Subjects (a Non-blinded, Parallel Group Study of Phase I)
Brief Title: Pharmacokinetics and Pharmacodynamics of BI 1356 in Subjects With Different Degrees of Liver Impairment as Compared to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1218.27
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — Linagliptin

ARMS (4):
- BI 1356 - healthy subjects (Experimental)
  Interventions: Drug: BI 1356
- BI 1356 - mild liver impairment (Experimental)
  Interventions: Drug: BI 1356
- BI 1356 - moderate liver impairment (Experimental)
  Interventions: Drug: BI 1356
- BI 1356 - severe liver impairment (Experimental)
  Interventions: Drug: BI 1356

INTERVENTIONS:
Drug: BI 1356

SUMMARY:
To investigate the influence of mild, moderate, and severe liver impairment on the pharmacokinetics and pharmacodynamics of linagliptin in comparison with a control group with normal hepatic function after single or multiple oral administration of 5 mg linagliptin tablets

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatic impairment determined by results of screening classified as mild (Child-Pugh class A, score 6 points), moderate (Child-Pugh class B, score 7 to 9 points) or severe (Child-Pugh class C, score 10 to 15 points)
* Healthy males and females based on a complete medical history, including physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Subjects in the respective groups were matched with regard to age (±10 years), weight (±20%) and gender
* Age 18 to 70 years, inclusive
* Body mass index 18.5 to 29.9 kg/m2, inclusive
* Creatinine clearance ≥80 mL/min (except for patients with severe hepatic impairment, see exclusion criteria) according to Cockroft & Gault
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice and local legislation

Exclusion Criteria:

Exclusion criteria for all subjects

* Surgery of the gastrointestinal tract (except appendectomy and oesophageal varices)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders (except hepatoportal encephalopathy)
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections (except non-progressive chronic hepatitis not being in a progressive state)
* History of relevant allergy or hypersensitivity (including allergy to study drug or its excipients)
* Use of drugs which might reasonably influence the results of the trial or prolong the QT or QTc intervals (based on the knowledge at the time of preparing the Clinical Trial Protocol) within 10 days prior to study drug administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to study drug administration or during the trial
* Smoking (more than 10 cigarettes, 3 cigars, or 3 pipes per day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (>100 mL within 4 weeks prior to study drug administration or during the trial)
* Excessive physical activities (within 1 week prior to study drug administration or during the trial)
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT or QTc intervals (e.g. repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for torsade de pointes such as heart failure, severe hypokalemia (<3.0 mmol/L), family history of long QT syndrome

Additional/modified exclusion criteria for healthy volunteers

* Any finding of the medical examination (including BP, PR, and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Intake of drugs with a long half-life (>24 h) within 1 month or less than 10 half-lives of the respective drug prior to study drug administration or during the trial
* Any laboratory value outside the reference range of clinical relevance

Additional/modified exclusion criteria for patients with hepatic impairment

* Decompensated gastrointestinal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
* Patients with severe liver impairment (Child-Pugh C): Severe concurrent renal dysfunction (e.g. due to hepatorenal syndrome) and a creatinine clearance <40mL/min
* Intake of drugs with a long half-life (>24 h) within 1 month or less than 10 half-lives of the respective drug prior to study drug administration or during the trial and intake of metformin; drugs taken for treatment of the underlying disease are excluded
* Any laboratory value outside the reference range that is of clinical relevance, except for parameters related to liver impairment (e.g. albumin, bilirubin, enzymes) and liver function tests according to Child-Pugh classification

Additional exclusion criteria for female subjects

* Pregnancy or intention to become pregnant within 2 months of study completion
* Positive pregnancy test
* Lack of adequate contraception (e.g. sterilisation, intrauterine device) or have not been using a barrier method of contraception for at least 3 months prior to the study
* Unwillingness or inability to use a reliable method of barrier contraception (e.g. diaphragm with spermicidal cream or jelly or condoms with spermicidal foam), during the study and up to 2 months after completion or termination of the trial
* Unwillingness of partner to use condoms
* Lactation period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration time curve of the analyte in plasma over the time interval from 0 to 24 h after the last dose at steady state) for healthy patients and patients with mild and moderate liver impairment | up to day 12
Cmax,ss (maximum concentration of the analyte in plasma at steady state) for healthy patients and patients with mild and moderate liver impairment | up to day 12
AUC0-24 (area under the concentration time curve of the analyte in plasma over the time interval from 0 to 24 h after the first dose) for patients with severe liver impairment | up to 24 hours after drug administration
Cmax (maximum concentration of the analyte in plasma) for patients with severe liver impairment | up to day 6

SECONDARY OUTCOMES:
Plasma protein binding | up to day 12
Model-derived AUCτ,ss for patients with severe liver impairment | up to day 6
Model-derived Cmax,ss for patients with severe liver impairment | up to day 6
Plasma dipeptidyl peptidase-4 (DPP-4) activity | up to day 6
Plasma DPP-4 concentration | Day 1 (Baseline)
Number of patients with adverse events | up to 47 days
Number of patients with clinically significant changes in vital signs (Blood Pressure (BP), Pulse Rate (PR)) | Baseline, up to day 19
Number of patients with clinically relevant findings in 12-lead electrocardiogram (ECG) | Baseline, up to day 19
Number of patients with clinically relevant findings in clinical laboratory tests | Baseline, up to day 19
Assessment of tolerability by investigator on a 4-point scale | day 19
tmax(ss) (time from last dose to maximum concentration of the analyte in plasma after single dose/at steady state) for healthy patients and patients with mild and moderate liver impairment | up to day 12
C24(ss) (concentration of the analyte in plasma at steady state after administration of the first or last dose at the end of the dosing interval) for healthy patients and patients with mild and moderate liver impairment | up to day 12
λz(ss) (terminal rate constant in plasma after single dose/at steady state) for healthy patients and patients with mild and moderate liver impairment | up to day 12
t1/2(ss) (terminal half-life of the analyte in plasma after single dose/at steady state) for healthy patients and patients with mild and moderate liver impairment | up to day 12
MRTpo(ss) (mean residence time of the analyte in the body after oral administration after single dose/at steady state) for healthy patients and patients with mild and moderate liver impairment | up to day 12
CL/F(ss) (apparent clearance of the analyte in the plasma after extravascular administration after single dose/at steady state) for healthy patients and patients with mild and moderate liver impairment | up to day 12
Vz/F(ss) (apparent volume of distribution during the terminal phase λz following extravascular administration after single dose/at steady state) for healthy patients and patients with mild and moderate liver impairment | up to day 12
AUC0-24 (area under the concentration time curve of the analyte in plasma over the time interval from 0 extrapolated to 24 h after the first dose for multiple dose groups) for healthy patients and patients with mild and moderate liver impairment | up to 24 hours after the first dose
Cmax (maximum concentration of the analyte in plasma after the first dose in multiple dose groups) for healthy patients and patients with mild and moderate liver impairment | up to day 12
%AUCtz-∞ (percentage of area under the concentration-time curve of the analyte in plasma over the time interval from the time of the last quantifiable data point extrapolated to infinity after single dose) in patients with severe liver impairment | up to day 6
AUC0-∞ (area under the concentration time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity after single dose in patients with severe liver impairment) | up to day 6
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point after single dose in patients with severe liver impairment) | up to day 6